CLINICAL TRIAL: NCT02588885
Title: Restoring Emotional, Sexual, and Physical Empowerment Through CBT & Trauma-sensitive Care: A Chronic Pelvic Pain Intervention
Acronym: RESPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15050501-IRB01
Record Dates: First submitted 2015-09-24; First posted 2015-10-28 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Pelvic Pain; Stress Disorders, Traumatic
Keywords: physical therapy; psychotherapy; dysfunctional sexual behavior; pelvic pain; posttraumatic stress; PTSD; chronic pain
MeSH Terms: conditions — Pelvic Pain; Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trauma-sensitive Care (Experimental): Participants will attend 7, one-hour psychotherapy sessions, which will be concurrent with trauma-sensitive care at physical therapy appointments.
  Interventions: Behavioral: Trauma-sensitive Care

INTERVENTIONS:
Behavioral: Trauma-sensitive Care — Psychological intervention
  1. education
  2. empowerment
  3. desensitization
  4. relaxation tools
  Physical therapy intervention
  1. techniques to address muscular tension
  2. empowerment
  3. comfort
  4. encouragement of trauma-related coping skills

SUMMARY:
This project will develop and preliminarily examine RESPECT, a trauma-sensitive psychological and physical therapy intervention to treat chronic pelvic pain, posttraumatic stress symptoms (PTS), and dysfunctional sexual behavior among women with sexual abuse histories. Patients will be recruited after being referred to pelvic floor physical therapy for treatment of chronic pelvic pain. Participants will complete seven sessions of individual cognitive behavioral psychotherapy. Physical therapy will be provided by clinicians who have been trained in trauma-sensitive treatment techniques. Treatment acceptability and outcomes will be assessed at baseline, mid intervention, post-intervention and follow-up via self-report measures. The RESPECT protocol is expected to be feasible to implement among sexual abuse survivors and to be well liked by patients. RESPECT is expected to reduce chronic pelvic pain, PTS, dysfunctional sexual behavior, treatment avoidance.

DETAILED DESCRIPTION:
This project will develop and preliminarily examine RESPECT, a trauma-sensitive psychological and physical therapy intervention to treat chronic pelvic pain, posttraumatic stress symptoms (PTS), and dysfunctional sexual behavior among women with sexual abuse histories. Chronic pelvic pain disorders are highly prevalent in the U.S., affecting between 10-21% of premenopausal women at some time in their lives. Chronic pelvic pain is associated with dyspareunia, depression, anxiety, relationship distress, functional impairment and poor quality of life. History of sexual abuse is associated with development of chronic pelvic pain and with the severity of psychological distress and functional impairment among chronic pain patients.

Unfortunately, frontline chronic pelvic pain treatments such as physical therapy and pain-specific psychological interventions fail to address sexual trauma. Standard physical therapy may actually trigger trauma related symptoms because it involves invasive techniques including internal digital palpation of pelvic floor muscles and the use of vaginal dilators. Neglecting trauma in chronic pelvic pain treatment could contribute to poor treatment outcomes, low adherence, and drop out. RESPECT's trauma-sensitive psychological intervention will teach women skills to cope with PTS, pain, sexual dysfunction, and discomfort during physical therapy. RESPECT's trauma-sensitive physical therapy intervention will more sensitively apply the invasive aspects of treatment and reinforce women's use of trauma-related coping skills learned in the psychological intervention. RESPECT is predicted to decrease chronic pelvic pain, PTS, dysfunctional sexual behavior, treatment avoidance.

Study Aims

1. Develop a multi-level trauma-sensitive (psychological and physical therapy) chronic pelvic pain intervention for inner-city women with histories of sexual abuse and PTS symptoms.
2. Examine the feasibility of RESPECT in treating this population.
3. Use a pilot open trial to examine the impact of RESPECT chronic pelvic pain, PTS, dysfunctional sexual behavior, treatment avoidance.

RESPECT's trauma-sensitive psychological intervention will 1) educate the patient about the relations between sexual abuse, PTS, and chronic pelvic pain 2) empower her by explaining that sexual abuse, chronic pelvic pain, and PTS are not her fault but she has the power to combat them 3) desensitize her to anxiety provoking components of the physical therapy intervention, and 4) teach her relaxation tools that she can use during physical therapy sessions, while practicing at-home physical therapy exercises, and to cope with pain more generally.

RESPECT's trauma-sensitive physical therapy intervention will 1) teach the patient techniques to address muscular tension that contributes to chronic pelvic pain 2) empower her by increasing her control over each phase of treatment (e.g., starting, stopping, expressing feelings and preferences) 3) comfort her by explaining that it is normal to experience discomfort during physical therapy treatment and 4) encourage her to use the trauma-related coping skills she learned in the psychotherapy component.

This initial project is intended to lead to a larger open trial that will examine not only treatment outcomes, but also the mechanisms of change (e.g., women's feeling of empowerment, decrease in PTS symptoms).

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* History of sexual abuse
* Premenopausal
* Chronic pelvic pain defined as pelvic pain with a duration of six months of at least a moderate severity

Exclusion Criteria:

* Not menstruating for reasons other than birth control
* Not currently receiving any current trauma-focused psychological treatment (i.e., prolonged exposure therapy, cognitive processing therapy, eye movement desensitization reprocessing)
* No current psychotic symptoms or current use of anti-psychotic medications
* No current suicidal ideation in the past month
* Not currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Chronic pelvic pain | 4 months
  Women will be asked to rate the severity of their pain during a variety of activities (e.g., pain at ovulation, pain while lifting) on a 10-point scale (0 = no pain, 10 = worst pain imaginable). Difference measured from pre to post intervention
Posttraumatic stress (PTS) - The 20-item PTSD Checklist for DSM-5 will be used to assess symptoms of Posttraumatic Stress Disorder. Items are rated on a 5-point Likert (scale with greater scores indicating more severe symptomatology | 4 months
  Difference from pre to post intervention
Sexual History FOrm | 4 months
  The SHF will be used to assess participants' sexual history. The Female Sexual Function Index will assess participant's sexual feelings and responses. Women are asked 37 questions. Difference measured from pre to post intervention
Treatment avoidance | 4 months
  Women's pelvic floor functioning will be assessed by collecting data from patient's medical records which is typically recorded as part of routine clinical practice. Difference measured from pre to post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Tirone, Ph.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush UMC Outpatient Physical Therapy Clinic, Chicago, Illinois, United States

REFERENCES:
- [Background] Armour C, Tsai J, Durham TA, Charak R, Biehn TL, Elhai JD, Pietrzak RH. Dimensional structure of DSM-5 posttraumatic stress symptoms: support for a hybrid Anhedonia and Externalizing Behaviors model. J Psychiatr Res. 2015 Feb;61:106-13. doi: 10.1016/j.jpsychires.2014.10.012. Epub 2014 Nov 22. PMID 25479765
- [Background] Chandler HK, Ciccone DS, Raphael KG. Localization of pain and self-reported rape in a female community sample. Pain Med. 2006 Jul-Aug;7(4):344-52. doi: 10.1111/j.1526-4637.2006.00185.x. PMID 16898946
- [Background] Jamieson DJ, Steege JF. The prevalence of dysmenorrhea, dyspareunia, pelvic pain, and irritable bowel syndrome in primary care practices. Obstet Gynecol. 1996 Jan;87(1):55-8. doi: 10.1016/0029-7844(95)00360-6. PMID 8532266
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Laumann EO, Paik A, Rosen RC. Sexual dysfunction in the United States: prevalence and predictors. JAMA. 1999 Feb 10;281(6):537-44. doi: 10.1001/jama.281.6.537. PMID 10022110
- [Background] Latthe P, Latthe M, Say L, Gulmezoglu M, Khan KS. WHO systematic review of prevalence of chronic pelvic pain: a neglected reproductive health morbidity. BMC Public Health. 2006 Jul 6;6:177. doi: 10.1186/1471-2458-6-177. PMID 16824213
- [Background] Lang AJ, Stein MB. An abbreviated PTSD checklist for use as a screening instrument in primary care. Behav Res Ther. 2005 May;43(5):585-94. doi: 10.1016/j.brat.2004.04.005. PMID 15865914
- [Background] Leclerc B, Bergeron S, Binik YM, Khalife S. History of sexual and physical abuse in women with dyspareunia: association with pain, psychosocial adjustment, and sexual functioning. J Sex Med. 2010 Feb;7(2 Pt 2):971-80. doi: 10.1111/j.1743-6109.2009.01581.x. Epub 2009 Nov 13. PMID 19912492
- [Background] Mark H, Bitzker K, Klapp BF, Rauchfuss M. Gynaecological symptoms associated with physical and sexual violence. J Psychosom Obstet Gynaecol. 2008 Sep;29(3):164-72. doi: 10.1080/01674820701832770. PMID 18821266
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159
- [Background] Mathias SD, Kuppermann M, Liberman RF, Lipschutz RC, Steege JF. Chronic pelvic pain: prevalence, health-related quality of life, and economic correlates. Obstet Gynecol. 1996 Mar;87(3):321-7. doi: 10.1016/0029-7844(95)00458-0. PMID 8598948
- [Background] McWilliams LA, Kowal J, Wilson KG. Development and evaluation of short forms of the Pain Catastrophizing Scale and the Pain Self-efficacy Questionnaire. Eur J Pain. 2015 Oct;19(9):1342-9. doi: 10.1002/ejp.665. Epub 2015 Mar 11. PMID 25766681
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Nicholson LM, Schwirian PM, Klein EG, Skybo T, Murray-Johnson L, Eneli I, Boettner B, French GM, Groner JA. Recruitment and retention strategies in longitudinal clinical studies with low-income populations. Contemp Clin Trials. 2011 May;32(3):353-62. doi: 10.1016/j.cct.2011.01.007. Epub 2011 Jan 27. PMID 21276876
- [Background] Osman A, Barrios FX, Kopper BA, Hauptmann W, Jones J, O'Neill E. Factor structure, reliability, and validity of the Pain Catastrophizing Scale. J Behav Med. 1997 Dec;20(6):589-605. doi: 10.1023/a:1025570508954. PMID 9429990
- [Background] Postma R, Bicanic I, van der Vaart H, Laan E. Pelvic floor muscle problems mediate sexual problems in young adult rape victims. J Sex Med. 2013 Aug;10(8):1978-87. doi: 10.1111/jsm.12196. Epub 2013 May 16. PMID 23679151
- [Background] Powers A, Fani N, Pallos A, Stevens J, Ressler KJ, Bradley B. Childhood abuse and the experience of pain in adulthood: the mediating effects of PTSD and emotion dysregulation on pain levels and pain-related functional impairment. Psychosomatics. 2014 Sep-Oct;55(5):491-9. doi: 10.1016/j.psym.2013.10.004. Epub 2013 Oct 23. PMID 24360527
- [Background] Rapaport MH, Clary C, Fayyad R, Endicott J. Quality-of-life impairment in depressive and anxiety disorders. Am J Psychiatry. 2005 Jun;162(6):1171-8. doi: 10.1176/appi.ajp.162.6.1171. PMID 15930066
- [Background] Reed BD, Haefner HK, Punch MR, Roth RS, Gorenflo DW, Gillespie BW. Psychosocial and sexual functioning in women with vulvodynia and chronic pelvic pain. A comparative evaluation. J Reprod Med. 2000 Aug;45(8):624-32. PMID 10986680
- [Background] Tripoli TM, Sato H, Sartori MG, de Araujo FF, Girao MJ, Schor E. Evaluation of quality of life and sexual satisfaction in women suffering from chronic pelvic pain with or without endometriosis. J Sex Med. 2011 Feb;8(2):497-503. doi: 10.1111/j.1743-6109.2010.01976.x. Epub 2010 Aug 16. PMID 20722779
- [Background] UyBico SJ, Pavel S, Gross CP. Recruiting vulnerable populations into research: a systematic review of recruitment interventions. J Gen Intern Med. 2007 Jun;22(6):852-63. doi: 10.1007/s11606-007-0126-3. Epub 2007 Mar 21. PMID 17375358
- [Background] Van Damme S, Crombez G, Bijttebier P, Goubert L, Van Houdenhove B. A confirmatory factor analysis of the Pain Catastrophizing Scale: invariant factor structure across clinical and non-clinical populations. Pain. 2002 Apr;96(3):319-324. doi: 10.1016/S0304-3959(01)00463-8. PMID 11973004
- [Background] Walker EA, Newman E, Koss M, Bernstein D. Does the study of victimization revictimize the victims? Gen Hosp Psychiatry. 1997 Nov;19(6):403-10. doi: 10.1016/s0163-8343(97)00061-3. PMID 9438184
- [Background] Zondervan K, Barlow DH. Epidemiology of chronic pelvic pain. Baillieres Best Pract Res Clin Obstet Gynaecol. 2000 Jun;14(3):403-14. doi: 10.1053/beog.1999.0083. PMID 10962634